CLINICAL TRIAL: NCT03623945
Title: Autoantibodies in Breast Cancer Detection
Acronym: ABCD
Status: Terminated | Type: Observational
Why Stopped: Study closed to enrollment and data and specimen collection due to lack of funding.
Sponsor: Sanford Health (Other)
Collaborators: Inanovate (Unknown)
Responsible Party: Sponsor
Other Study IDs: SH ABCD
Record Dates: First submitted 2018-07-26; First posted 2018-08-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Cohort A: Patients who have recently had an abnormal mammogram, followed by a breast biopsy and an initial diagnosis of Stage I, II, III or IV invasive breast cancer, will be invited to participate. Stage I, II and III participants will be further categorized into high-risk and low-risk. For the purposes of this study, participants with at least one of the following will be considered high-risk; any triple negative cancer, any grade III cancer, lymph node involvement, tumor greater than 2cm, or any patient receiving cytotoxic chemotherapy.
  Interventions: Other: Collection of blood
- Cohort B: Patients who have recently had an abnormal mammogram, followed by a breast biopsy and diagnosed with a benign but high-risk pathology, will be invited to participate. This includes, but is not limited to, atypical ductal hyperplasia, atypical lobular hyperplasia, ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), flat epithelia atypia or phylloides.
  Accrual to Cohort B is complete.
  Interventions: Other: Collection of blood
- Cohort C: Patients who have recently had an abnormal mammogram, followed by a breast biopsy and diagnosed with a benign tumor, will be invited to participate. This includes, but is not limited to, fibroadenoma, papilloma, fibrocystic changes and Pseudoangiomatous stromal hyperplasia (PASH). Accrual to Cohort C is complete
  Interventions: Other: Collection of blood
- Cohort D: Patients who have had a normal screening mammogram within the last 6 months will be invited to participate. Accrual to Cohort D is complete.
  Interventions: Other: Collection of blood
- Cohort E: Patients who have recently had an abnormal mammogram, followed by a breast biopsy and an initial diagnosis of Stage I, II, III invasive breast cancer.
  Patients who have recently had an abnormal mammogram, followed by a breast biopsy, and diagnosed with a benign but high-risk pathology.
  Cohort E has 3 sub-groups. For the purposes of this study, participants with a breast cancer will be categorized as E1-malignant high risk, of E2-malignant low risk.
  Patients who have recently had an abnormal mammogram, followed by a breast biopsy, and diagnosed with a benign but high-risk pathology, will be invited to participate.
  These patients will be considered E3-benign high-risk.
  Interventions: Other: Collection of blood

INTERVENTIONS:
Other: Collection of blood — Collection of blood only to look at circulating autoantibodies that recognize breast cancer proteins to potentially be used as a biosensor for identifying patients with increased risk of having breast cancer

SUMMARY:
Prospective, single-center study in women who have recently had an abnormal mammogram followed by a breast biopsy or women who have recently had a normal screening mammogram. We are no longer enrolling women who had normal Screening mammograms.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

All Cohorts:

* Women age 18 and older
* Understand and provide informed consent and HIPAA Authorization prior to initiation of any study-specific procedures

Cohort A:

* Recent abnormal mammogram followed by a breast biopsy
* Initial diagnosis of Stage I, II, III or IV invasive breast cancer

Cohort B:

* Recent abnormal mammogram followed by a breast biopsy
* Diagnosed benign breast tumor with high-risk pathology. This would include, but is not limited to, atypical ductal hyperplasia, atypical lobular hyperplasia, lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS), flat epithelia atypia and phylloides

Cohort C:

* Recent abnormal mammogram followed by a breast biopsy
* Diagnosed benign breast tumor. This would include, but is not limited to, fibroadenoma, papilloma, fibrocystic changes, and Pseudoangiomatous stromal hyperplasia (PASH)

Cohort D:

• Normal screening mammogram within the last 6 months

Exclusion Criteria:

* All Cohorts:

  * Men.
  * Unable or unwilling to give written informed consent

Cohort A:

• History of cancer other than non-melanoma basal or squamous cell skin carcinoma, ductal carcinoma in situ (DCIS) and cervical carcinoma in situ.

Cohort B:

• History of cancer other than non-melanoma basal or squamous cell skin carcinoma and cervical carcinoma in situ.

Cohort C:

• History of cancer other than non-melanoma basal or squamous cell skin carcinoma and cervical carcinoma in situ.

Cohort D:

* History of cancer other than non-melanoma basal or squamous cell skin carcinoma and cervical carcinoma in situ.
* History of or current autoimmune disease including but not limited to Sjogrens Syndrome, Systemic Sclerosis (SSc), Scleroderma (Scl) and Dermatomyositis, Systemic Lupus Erythematosus, Multiple Sclerosis, Type I Diabetes, Rheumatoid Arthritis
* History of abnormal mammogram

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients only
Study Population: Women who have recently had an abnormal mammogram followed by a breast biopsy or women who have recently had a normal screening mammogram.
  The study team will enroll approximately 1,550 participants at Sanford Health in Sioux Falls, SD and Fargo, ND. Cohort A= 300 participants, Cohort B= 250 participants, Cohort C= 500 participants and Cohort D= 500 participants.
Sampling Method: Non-Probability Sample
Enrollment: 1279 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Autoantibodies for breast cancer diagnosis | 5 years
  The data from Phase I will be tested and validated with newly diagnosed BCa patient samples from Cohort A, and age-matched healthy controls taken from Cohort D, and a risk score will be developed based on a composite of autoantibodies for breast cancer diagnosis. A Cox Proportional Hazards (PH) Regression will be used to analyze a case-cohort study design to validate the risk score by identifying breast cancer cases from those cases in Cohorts B, C and D.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Watson, MD, Principal Investigator — Sanford Health
Locations (2):
- United States (2):
  - Sanford Health, Fargo, North Dakota
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data